CLINICAL TRIAL: NCT05081947
Title: Assessing the Acceptability and Feasibility of COMPASS, a Transdiagnostic Web-based Intervention for the Management of Depression and Anxiety in Long-term Conditions, in Community-based Heart Failure Patients
Brief Title: Assessing the Acceptability and Feasibility of COMPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 288961
Record Dates: First submitted 2021-09-23; First posted 2021-10-18 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2021-09

CONDITIONS: Heart Failure; Depression; Anxiety
MeSH Terms: conditions — Heart Failure; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heart failure patients (Other): patients will try the Compass intervention
  Interventions: Behavioral: COMPASS

INTERVENTIONS:
Behavioral: COMPASS — COMPASS is a web-based intervention (online CBT program) that was developed for managing illness-related anxiety and depression in patients with long-term conditions (LTC) (https://compass-ltc.org/). An example of the patient login page can be viewed here: www.compass-southwark.co.uk. COMPASS aims to support people in managing the challenges of living with a long-term condition. COMPASS is based on research which shows the benefit of combining mental and physical healthcare. The proposed COMPASS program consists of 11 online sessions for patients to work through over approximately 12 weeks. The sessions can be worked through in any order the patient would like. The sessions are split into four quadrants - North, East, South and West - which explore different elements of managing the LTC challenges that were identified from the evidence-based systematic review. Sessions contain information, interactive tasks, goal setting and patient stories.

SUMMARY:
Heart failure (HF) is a complex clinical syndrome characterized by the inability of the heart to pump an adequate amount of blood. Heart failure affects patients' ability to carry out even simple activities of daily living and therefore has a negative psychological impact. Many studies reported that anxiety and depression are prevalent among HF patients and it is being associated with high morbidity, mortality and costs. Community HF patients who are diagnosed with depression are usually referred for Improving Access for Psychological Therapies (IAPT). The IAPT services have long waiting lists and many patients in the community still do not have access to IAPT. IAPT (2017) found web-based interventions for psychological therapies for emotional disorders such as depression and anxiety to be as effective as the traditional interventions and yielded positive mental health outcomes.

In this current study, the feasibility and acceptability of the proposed COMPASS web-based intervention will be examined. COMPASS is a web-based therapy (online CBT program) designed for the management of depression and anxiety for patients with long term conditions such as heart failure.

This study will be conducted into three parts and mainly include one-to-one interviews. First, the researcher will use an approach called "think aloud" which is a specific type of interview that allows us to observe the participant while using the proposed COMPASS online using Microsoft Teams. The participant will be asked to log into the COMPASS website and talk to the researcher continuously as possible about what they are thinking or what comes into their mind as they are using the COMPASS website. Following this interview, the researcher will ask the participant to use COMPASS from any internet-connected device for four weeks with weekly follow-up telephone calls. One month after the completion of COMPASS, the researcher will interview the participants.

DETAILED DESCRIPTION:
Heart failure (HF) is the inability of the heart muscle to pump enough blood to meet the body's blood and oxygen requirements. The European Society of Cardiology (ESC) described HF as a clinical syndrome resulting from the reduced cardiac output that may be accompanied with high intracardiac pressure during rest or with stress. It is characterized by shortness of breath, fatigue and limited exercise tolerance. The prevalence of HF is increasing worldwide, and HF cases increased by 23% in the United Kingdom (UK) from 2002 to 2014. In the year 2017-2018 in England, 500,000 people were diagnosed with heart failure. According to hospital diagnoses in the UK, there were up to 920,000 people living with HF. Many HF patients develop anxiety and depression due to the pathological similarities in both conditions. The prevalence of major in depression in HF is reported to be around 20-40% that is more than the reported prevalence in the normal population.

The National Institute for Health and Care Excellence (NICE) guidelines on HF emphasized the importance of treating depression in HF but there were no specific treatment options for HF recommended in the document. The ESC HF recommended initiating depression treatment for all HF patients using psychosocial interventions, pharmacological therapy or exercise training. In Southwark and Lambeth Boroughs, the community-based HF patients who are diagnosed with depression are usually referred for psychological treatment such as Improving Access for Psychological Therapies (IAPT) or 3 Dimensions for Long Term Conditions (3DLC). The type of treatment depends on the severity of their depression and the extent to which depression is affecting clients' self-management of HF. So, for persistent and mild to moderate depression or if the depression is not related to HF, the patients will be referred to IAPT for treatment. While, for moderately severe to severe depression and whose depression affects their management of HF, patients will be seen by the team of 3DLC. The IAPT services have long waiting lists and many patients in the community with anxiety and depression still do not have access to IAPT. The impact of the Covid-19 pandemic has increased the burden further on IAPTS services.

This current study builds on our phase 2 study (268951) which is currently using online focus group with community HF nurses (n=5) and qualitative telephone/online interviews with community-based HF patients (n=8) to examine their views and experiences in managing depression and anxiety in the primary setting, and whether the proposed COMPASS, a web-based intervention, can be used for managing depression and anxiety in community-based HF patients. The findings from phase 2 study will be analysed to identify patients' perspectives and readiness to use the web-based COMPASS intervention for managing anxiety and depression in HF.

In this study (phase 3), the feasibility and acceptability of the proposed COMPASS web-based intervention will be examined with community-based HF patients. Web-based interventions such as COMPASS are programs or applications that can be accessed through the website. They are usually developed to change health behaviour, provide education, monitor symptoms or deliver interventions. Barak et al. (2009) defined a web-based intervention as programs that are primarily self-guided and that are delivered online for people requiring health and mental health-related support. These interventions aim to improve knowledge or create awareness through the delivery of health-related content in an interactive web-based program.

IAPT (2017) found web-based interventions for psychological therapies for emotional disorders such as depression and anxiety to be as effective as the traditional interventions and yielded positive mental health outcomes. Web-based interventions allow the intervention to be delivered through a patient-centred approach that is strengthened by the support of trained therapist. With the rapid advancement in technology and the widespread use of the internet, web-based interventions have grown in popularity as they are seen as cost-effective, and easily accessible from a patient perspective (Murray, 2012). Web-based interventions aim to improve self-management skills of patients with chronic diseases such as cardiovascular diseases, diabetes, and arthritis. Web-based interventions for chronic cardiac conditions were reported to be cost-effective, easily accessible by participants through different devices (laptops, smartphones or computers), confidential, non-stigmatizing and acceptable. Patients can easily fit the web-based interventions into their daily life, and it can be easily approached by HF patients.

COMPASS is a web-based intervention (online CBT program) that was developed for managing illness-related anxiety and depression in patients with long-term conditions. COMPASS aims to support people in managing the challenges of living with a long-term condition. COMPASS is based on research that shows the benefit of combining mental and physical healthcare. COMPASS was developed by a team of experienced health psychology researchers and practitioners at King's College London. The structure and content of COMPASS are based on a systematic review to identify mechanisms of action which trigger and sustain symptoms of depression and/or anxiety in the context of LTCs. COMPASS is tailored to gain an understanding of the difficulties that LTC patients experience and provide information and tools on how to manage these.

COMPASS is different from other web-based talking therapy because it:

* is tailored to treat low mood and anxiety in the context of living with one or more long-term conditions.
* uses the latest research evidence to identify mechanisms known to trigger and sustain symptoms of low mood and anxiety in people with long-term conditions. These mechanisms are then targeted in the program.
* has been co-developed by people with long-term conditions to improve its acceptability, utility and ease of use.

The proposed COMPASS program consists of 11 online sessions for patients to work through over approximately 12 weeks. The sessions can be worked through in any order the patient would like. The sessions are split into four quadrants - North, East, South and West - which explore different elements of managing the LTC challenges that were identified from the evidence-based systematic review. Sessions contain information, interactive tasks, goal setting and patient stories.

If the proposed COMPASS is found to be applicable to use in HF, this will help patients who are considered vulnerable and are shielding from, for example, the COVID-19 outbreak. During the pandemic, patients were unable to attend for psychological therapies that were conducted face to face, thus the use of COMPASS will assist in delivering the psychological intervention for a large number of patients anywhere and at any time. In this study, the acceptability and feasibility of COMPASS as a web-based intervention during the Covid-19 pandemic will be also explored as a virtual therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

* Community-based HF patients from community HF service and outpatient department with depression and anxiety related to their HF will be invited to participate in the study. The inclusion criteria include:

  * Adults over 18 years of age;
  * community-based HF patients capable of providing written/verbal informed consent;
  * Community-based HF patients with mild to moderately-severe depression (using PHQ-9) with/without anxiety symptoms related to their HF;
  * community-based HF patients who are not engaging in any psychological treatment at the time of recruitment;
  * Is fluent in the English language so can fully respond to verbal and written material; and
  * Has access to the internet and has an electronic device (i.e. computer, laptop etc).

Exclusion Criteria:

* The exclusion criteria include community-based HF patients:

  * With severe depression validated by PHQ-9 score (> 19) as assessed by the researcher;
  * who are receiving or engaging in other psychological treatment for anxiety and depression;
  * have active suicidal ideation if reported during the assessment with the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
COMPASS Acceptability and feasibility as measured by Treatment Acceptability/Adherence Scale (TAAS) and interviews | This will be measured at first Think aloud Interview (immediately after first use of compass)
  TAAS is a 10 items self-reported scale rated on a 7- point Likert scale. Possible scores can range from 10 to 70, and higher scores are indicative of higher acceptability of treatment and greater anticipated ability to adhere to it.
COMPASS Acceptability and feasibility as measured by Treatment Acceptability/Adherence Scale (TAAS) and interviews | This will be measured second time at week 4 follow up post Compass use
  TAAS is a 10 items self-reported scale rated on a 7- point Likert scale. Possible scores can range from 10 to 70, and higher scores are indicative of higher acceptability of treatment and greater anticipated ability to adhere to it.
Treatment usability using the System Usability Scale (SUS) | This will be measured at weekly basis at each session after using compass and for a total of 4 weeks
  SUS scores have a range of 0 to 100. SUS yields a single number representing a composite measure of the overall usability of the intervention being used.

SECONDARY OUTCOMES:
changes in depression scores as measured by Patient Health Questionnaire-9 (PHQ-9) | every 2 weeks after using compass. First it will be measures at baseline (before compass) and then every 2 weeks.
  The score ranges from 0-27 with highre scores indicating sever deprssion
changes in anxiety score as measured by Generalised Anxoety Disorder-7 (GAD-7) | every 2 weeks after using compass. First it will be measures at baseline (before compass) and then every 2 weeks.
  The score ranges from 0-21 with highre scores indicating sever anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Failure Community Service, London, Westminester, United Kingdom

IPD SHARING:
Plan to Share IPD: No